CLINICAL TRIAL: NCT02499705
Title: The Effect of Artificial Sweeteners (AFS) on Sweetness Sensitivity, Preference and Brain Response in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Prematurely unblinded based on outcome in other trial. 2 out of 3 particpants in one arm had clinically elevated fasting insulin. Adverse event was reported.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 1409014612
Record Dates: First submitted 2015-01-06; First posted 2015-07-16 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — trichlorosucrose; Sucrose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sucralose (Experimental): Flavored beverage with sucralose.
  Interventions: Dietary Supplement: Sucralose
- Sucrose (Experimental): Flavored beverage with sucrose.
  Interventions: Dietary Supplement: Sucrose
- Sucralose + maltodextrin (Experimental): Flavored beverage with Splenda + maltodextrin .
  Interventions: Dietary Supplement: Sucralose + maltodextrin

INTERVENTIONS:
Dietary Supplement: Sucralose — 2 packets
  Arms: Sucralose
Dietary Supplement: Sucrose — equisweet to sucralose
  Arms: Sucrose
Dietary Supplement: Sucralose + maltodextrin — sucralose plus equicaloric (to sucrose) maltodextrin
  Arms: Sucralose + maltodextrin

SUMMARY:
The purpose of this study is to investigate the effects of dietary exposure to artificial sweeteners on taste sensitivity, preference and brain response in adolescents using fMRI, psychophysical measures, and questionnaires. The investigators hypothesize that dietary exposure to artificial sweeteners (sucralose) will decrease sensitivity to taste, shift preference of sweet and savory taste to a higher dose, and reduce brain response in amygdala to sweet taste compared to sucrose.

DETAILED DESCRIPTION:
We aim to identify neural factors that contribute to taste intensity perception in humans and to determine environmental mechanisms that contribute to variation in taste sensitivity. Significant controversy surrounds the possibility that consumption of artificial sweeteners (AFS) leads to weight gain. Given that the five FDA approved AFSs are found in thousands of foods (Yang 2010) this marks a clear and significant gap in knowledge. Our preliminary data demonstrate a 3-fold decrease in sweet taste sensitivity following consumption of a beverage sweetened with two packets of Splenda for just 10 days. These data provide strong evidence that repeated exposure to sucralose reduces perception of sweet taste intensity, most likely by down-regulation of the sweet taste receptor. Adolescents may be more sensitive to exposure to AFS because of changes in metabolism during this period of development. Physiologic insulin resistance occurs during adolescence (Moran, Jacobs et al. 1999); this change in insulin sensitivity may predispose adolescents to greater impairments in sweet taste intensity by altering the relationship between sweet taste and post-ingestive reward, as suggested by the Davidson and Swithers model (Davidson and Swithers 2004). Therefore, it is imperative that we gain a greater understanding of the physiological consequences of AFS use in adolescents, since alterations in sweet taste perception, metabolism and brain reward that occur in response to AFS exposure may promote weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Fluent in English
* Right handed
* 13-17 years old

Exclusion Criteria:

* History of oral nerve damage, presence of known taste or smell disorder, food allergies or sensitivities (for example nuts, lactose, artificial sweeteners), history of CNS disease, diabetes, history of DSM-IV major psychiatric disorder, including alcohol and substance abuse, chronic use of medication that may affect taste, conditions that may interefere with gustatory or olfactory perception (colds, seasonal allergies, recent smoking history), aberrant stimulus ratings, contra-indication for fMRI, uncomfortable swallowing in supine position, discomfort or anxiety associated with insertion an intravenous catheter, regular artificial sweetener use.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Ratings of taste sensitivity | on average 2 weeks
  At baseline and after on average 2 weeks, subjects will rate intensity of sucrose, sucralose, mono potassium glutamate, sodium chloride and citric acid using the General Labeled Magnitude Scale (gLMS). It is a vertical line with quasi-logarithmic spaced labels that start at the bottom with 'barely detectable' to 'strongest imaginable' at the top, recoded to 0-100.

SECONDARY OUTCOMES:
Insulin resistance and GLP-1 | on average 2 weeks
  We will draw a blood sample to assess glucose, insulin and GLP-1
Ad libitum food intake | on average 2 weeks
  Subject is offered milk and cereal and asked to consume as much as they want. The amount consumed is measured in weight and converted to calories.
percent signal change of brain response in reward and gustatory areas to taste stimuli | on average 2 weeks
  brain response in reward and gustatory areas to sucrose, mono potassium glutamate, sodium chloride and citric acid (in percent signal change).

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, PhD, Principal Investigator — The John B. Pierce Laboratory/Yale University
Locations (1):
- The John B. Pierce Laboratory, New Haven, Connecticut, United States